CLINICAL TRIAL: NCT00445601
Title: A Phase III Blinded Study of Immediate Post TURBT Instillation of Gemcitabine Versus Saline in Patients With Newly Diagnosed or Occasionally Recurring Grade I/II Superficial Bladder Cancer
Brief Title: S0337, Gemcitabine After Surgery in Treating Patients With Newly Diagnosed or Recurrent Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDR0000534235; S0337 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Results first posted 2018-04-24 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Bladder Cancer
Keywords: transitional cell carcinoma of the bladder; stage 0 bladder cancer; stage I bladder cancer; recurrent bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Patients receive intravesical gemcitabine hydrochloride over 1 hour.
  Interventions: Drug: gemcitabine hydrochloride
- Arm II (Placebo Comparator): Patients receive intravesical placebo over 1 hour.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given intravesically
  Arms: Arm I
Other: placebo — Given intravesically
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving gemcitabine directly into the bladder after surgery may kill more tumor cells. It is not yet known whether giving gemcitabine directly into the bladder is more effective than a placebo in treating bladder cancer.

PURPOSE: This randomized phase III trial is studying gemcitabine to see how well it works when given directly into the bladder compared with a placebo after surgery in treating patients with newly diagnosed or recurrent bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of a single intravesical instillation of gemcitabine hydrochloride vs placebo immediately after transurethral resection of the bladder tumor (TURBT) in preventing recurrence at 2 years in patients with grade 1 or 2 superficial transitional cell cancer of the bladder.

Secondary

* Compare whether a single instillation of intravesical gemcitabine hydrochloride can improve the time to progression to muscle invasive disease vs placebo in these patients.
* Compare the qualitative and quantitative toxicities of these regimens in these patients.
* Compare whether treatment with post-TURBT intravesical instillation of gemcitabine vs placebo results in reduced long-term morbidity in patients, as defined by requirement for fewer TURBTs, courses of traditional intravesical therapies, and surveillance cystoscopies over 4 years.

Tertiary

* Assess whether performing a combination of molecular and/or cytologic diagnostic marker tests, including NMP-22 Bladder Chek and BTA Stat every 3 months, can predict recurrence as accurately as cystoscopy alone in these patients.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients are stratified according to disease status (first occurrence vs recurrent disease) and number of tumor sites (1 vs ≥ 2). Patients are randomized to 1 of 2 treatment arms.

All patients undergo transurethral resection of the bladder tumor. Within 3 hours, patients receive intravesical therapy according to their randomized arm.

* Arm I: Patients receive intravesical gemcitabine hydrochloride over 1 hour.
* Arm II: Patients receive intravesical placebo over 1 hour. Urine is collected at baseline and then every 3 months for 2 years for research studies including the NMP-22 Bladder Chek and BTA Stat test.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 340 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of newly diagnosed or recurrent transitional cell bladder cancer meeting the following criteria:

  * Ta or T1 primary tumor
  * Grade 1 or 2 disease
* No more than 2 recurrences (except for index tumor) within the 18 months prior to the index tumor's transurethral resection of the bladder tumor (TURBT)

  * Index tumor post-TURBT must meet the following criteria:

    * Ta or T1 tumor without any prior tumor in situ, grade 3 (high grade) disease within 2 years prior to index tumor TURBT, or invasion of the muscularis propria (stage ≥ T2)
    * Grade 1 or 2 disease (similar to papillary urothelial neoplasm of low malignant potential and low-grade bladder cancer)
* Not a candidate for a therapy other than TURBT (e.g., a series of instillations of intravesical immunotherapy [e.g., BCG] or intravesical chemotherapy, or cystectomy or partial cystectomy)
* Negative upper tract imaging studies within 1 year (365 days) prior to study entry

  * Imaging studies may be performed after registration provided it is done prior to TURBT on the day of treatment
* No urothelial cancer of the prostate or more distal urethra (or urethra at all in women) as assessed by endoscopy
* Must have a negative urine culture (less than or equal to 10,000 col/mL, mixed flora-likely contamination) OR negative urine analysis for infection AND negative nitrates on reagent strip, ≤ 10 white blood cell count (WBC)/high-power field, and no rods or organisms on examination of spun urine sediment OR an automated or visual reagent strip urinalysis that is negative for leukocytes and nitrates within the past 28 days
* TURBT planned within the next 28 days and planned treatment within 3 hours after TURBT

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior malignancy except for any of the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated stage I or II cancer from which patient is in complete remission
  * Any other cancer from which patient has been disease-free for 3 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 145 days since prior intravesical therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2007-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward M. Messing, MD, FACS, Study Chair — James P. Wilmot Cancer Center; Deepak M. Sahasrabudhe, MD, Study Chair — James P. Wilmot Cancer Center; Theresa M. Koppie, MD, Study Chair — Oregon Health and Science University; David P. Wood, MD, Study Chair — Beaumont Physician Partners
Locations (70):
- United States (70):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Urology Center of Colorado, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - St. Joseph Regional Medical Center, Lewiston, Idaho
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - St. Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Hutchinson Hospital Corporation, Hutchinson, Kansas
  - Kansas City Cancer Centers - West, Kansas City, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - Mount Carmel Regional Cancer Center, Pittsburg, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Kansas City Cancer Center - Shawnee Mission, Shawnee Mission, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Kansas City Cancer Centers - East, Lee's Summit, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Bay Area Hospital, Coos Bay, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - Overlake Cancer Center at Overlake Hospital Medical Center, Bellevue, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington

REFERENCES:
- [Derived] Corsi NJ, Messing EM, Sood A, Keeley J, Bronkema C, Rakic N, Jamil M, Dalela D, Arora S, Piontkowski AJ, Majdalany SE, Butaney M, Rakic I, Li P, Menon M, Rogers CG, Abdollah F. Risk-Based Assessment Of the Impact Of Intravesical Therapy on Recurrence-Free Survival Rate Following Resection of Suspected Low-grade, Non-muscle-invasive Bladder Cancer (NMIBC): A Southwest Oncology Groups (SWOG) S0337 Posthoc Analysis. Clin Genitourin Cancer. 2022 Dec;20(6):e498-e505. doi: 10.1016/j.clgc.2022.06.015. Epub 2022 Jun 25. PMID 35871040
- [Derived] Messing EM, Tangen CM, Lerner SP, Sahasrabudhe DM, Koppie TM, Wood DP Jr, Mack PC, Svatek RS, Evans CP, Hafez KS, Culkin DJ, Brand TC, Karsh LI, Holzbeierlein JM, Wilson SS, Wu G, Plets M, Vogelzang NJ, Thompson IM Jr. Effect of Intravesical Instillation of Gemcitabine vs Saline Immediately Following Resection of Suspected Low-Grade Non-Muscle-Invasive Bladder Cancer on Tumor Recurrence: SWOG S0337 Randomized Clinical Trial. JAMA. 2018 May 8;319(18):1880-1888. doi: 10.1001/jama.2018.4657. PMID 29801011
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Patients receive intravesical gemcitabine hydrochloride over 1 hour post-TURBT.
  gemcitabine hydrochloride: Given intravesically
- Arm II: Patients receive intravesical placebo over 1 hour post-TURBT.
  placebo: Given intravesically
Period: Overall Study
Arm/Group | Arm I | Arm II
Started (Randomized to Treatment Arm) | 201 | 205
Received TURBT | 190 | 193
Completed (Received Drug Instillation) | 168 | 177
Not Completed | 33 | 28
Not completed — Withdrawal by Subject | 11 | 11
Not completed — TURBT Complication | 12 | 8
Not completed — Incorrect Disease Status | 6 | 6
Not completed — Drug Delivery Issue | 2 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Death prior to TURBT | 0 | 1

BASELINE CHARACTERISTICS:
Population: All eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 201 | 205 | 406
Age, Continuous [Median (Full Range); unit: years] | 66 [38 to 97] | 66 [35 to 93] | 66 [35 to 97]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 24 | 62
  Male | 163 | 181 | 344
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 186 | 185 | 371
  Race: Black | 6 | 9 | 15
  Race: Asian | 4 | 5 | 9
  Race: Native American | 0 | 2 | 2
  Race: Unknown | 5 | 4 | 9
Occurence status [Count of Participants; unit: Participants]
  First Occurence | 128 | 128 | 256
  Recurrent | 66 | 77 | 143
  Unknown | 7 | 0 | 7
Number of tumors [Count of Participants; unit: Participants]
  1 | 135 | 140 | 275
  >= 2 | 66 | 65 | 131
Prior intravesical therapy [Count of Participants; unit: Participants]
  Yes | 39 | 39 | 78
  No | 162 | 166 | 328
Zubrod Performance Status [Count of Participants; unit: Participants] — Zubrod Performance Status Scale:
  0. Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  3. Capable of limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled; cannot carry on any self-care; totally confined to bed or chair.
  Participants
    0 | 157 | 165 | 322
    1 | 44 | 40 | 84
Smoking history [Count of Participants; unit: Participants]
  Current | 49 | 54 | 103
  Prior | 98 | 101 | 199
  Never | 54 | 46 | 100
  Unknown | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Disease Recurrence Rate
Description: Percentage of patients who experienced a recurrence of grade 1 or 2 superficial transitional cell cancer of the bladder between the date of registration and 24 months. Disease recurrence considered to occur at date of first observation of recurrent disease subsequently confirmed by biopsy. Patients without recurrence were censored at the time of their last cystoscopy.
Time Frame: Up to 2 Years
Population: Intent-to-Treat population
Measure: Number; unit: percentage of patients with recurrence
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 201 | 205
percentage of patients with recurrence | 27.86 | 40
Statistical Analysis 1: Comparison: Arm I vs Arm II; Test type: Superiority; p = 0.01, Log Rank; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.48 to 0.90]

2. Secondary Outcome: Rate of Progression to Muscle Invasive Disease at 4 Years
Description: From date of registration to date of diagnosis of progressive disease. Censor at date of last disease assessment for those without progression.
Time Frame: 4 years
Population: Intent-to-Treat Population
Measure: Number; unit: percentage of patients with progression
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 201 | 205
percentage of patients with progression | 2.49 | 4.39
Statistical Analysis 1: Comparison: Arm I vs Arm II; Test type: Superiority; p = 0.23, Log Rank; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.18 to 1.49]

3. Secondary Outcome: Compare Qualitative and Quantitative Toxicities Between the Treatment Arms
Description: Number of patients with Grade 3 through Grade 5 adverse events that are related to study drug
Time Frame: Up to 4 years after Transurethral Resection of Bladder Tumor (TURBT)
Population: All eligible patients who received instillation after TURBT and reported adverse events
Measure: Number; unit: Participants
Groups:
- Arm I: Gemcitabine: Patients receive intravesical gemcitabine hydrochloride over 1 hour post-TURBT.
- Arm II: Placebo: Patients receive intravesical placebo over 1 hour post -TURBT.
Arm/Group | Arm I: Gemcitabine | Arm II: Placebo
Number analyzed (Participants) | 165 | 174
Participants
  Bladder spasms | 0 | 1
  Hemorrhage, GU - Bladder | 1 | 0
  Hemorrhage, GU - Urinary NOS | 2 | 1
  Infection-Other (Specify) | 1 | 0
  Pain - Bladder | 0 | 1
  Pain - Urethra | 0 | 1
  Urinary frequency/urgency | 0 | 2

4. Secondary Outcome: Rate of Disease Worsening Over 2 Years
Description: Compare whether treatment with post-TURBT intravesical instillation of gemcitabine vs placebo results in reduced long-term morbidity in patients, as defined by requirement for fewer TURBTs, courses of traditional intravesical therapies, and surveillance cystoscopies over 4 years.
Time Frame: Up to 2 years
Population: TURBT data after patients stopped trial was not collected.
Arm/Group | Arm I: Gemcitabine | Arm II: Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 2 years
Description: Participants were monitored for toxicity at Week 1 and 2 after protocol treatment, with an additional assessment at Week 4 if any toxicities noted during the first two weeks. Patients were then monitored every 3 weeks for the first 2 years following protocol treatment, and then every 6 months for the following 2 years (up to 4 years).
Groups:
- Arm II: Placebo: Patients receive intravesical placebo over 1 hour post-TURBT.
Arm/Group | Arm I: Gemcitabine | Arm II: Placebo
All-Cause Mortality (participants affected / at risk) | 17/201 | 25/205
Serious Adverse Events (participants affected / at risk) | 7/165 | 5/174
Other Adverse Events (participants affected / at risk) | 60/165 | 58/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Gemcitabine (N=165) | Arm II: Placebo (N=174)
Cardiac General-Other (Cardiac disorders) | 1 | 0
Infection with unknown ANC - Blood (Infections and infestations) | 0 | 1
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 0 | 1
Infection-Other (Infections and infestations) | 1 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 | 0
Tumor flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 1 | 0
Vasovagal episode (Nervous system disorders) | 1 | 0
Hemorrhage, GU - Bladder (Renal and urinary disorders) | 2 | 0
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 0 | 1
Obstruction, GU - Bladder (Renal and urinary disorders) | 0 | 1
Obstruction, GU - Ureter (Renal and urinary disorders) | 1 | 0
Pain - Bladder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Gemcitabine (N=165) | Arm II: Placebo (N=174)
Nausea (Gastrointestinal disorders) | 11 | 3
Vomiting (Gastrointestinal disorders) | 9 | 1
Bladder spasms (Renal and urinary disorders) | 13 | 9
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 16 | 19
Pain - Bladder (Renal and urinary disorders) | 23 | 23
Urinary frequency/urgency (Renal and urinary disorders) | 25 | 25
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 9 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-10-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT00445601/Prot_SAP_ICF_000.pdf